CLINICAL TRIAL: NCT01633008
Title: Acceptance and Commitment Therapy for Adolescents and Adults With Neurofibromatosis Type 1 and Chronic Pain: A Pilot Study
Brief Title: Acceptance and Commitment Therapy for Adolescents and Young Adults With Neurofibromatosis and Chronic Pain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120155; 12-C-0155
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2017-01-10

CONDITIONS: Neurofibromatosis
Keywords: Modified Brief Pain Inventory; Quality of Life; Pain-Related Coping; Pain-Related Anxiety; Depression
MeSH Terms: conditions — Neurofibromatoses; Depression

ARMS (1):
- 1 (Experimental): Attend three 2-hour sessions held over two consecutive days
  Interventions: Behavioral: ACT Workshop

INTERVENTIONS:
Behavioral: ACT Workshop — The ACT workshops will consist of a patient program and a corresponding parent program, each focusing on helping participants cope with the patient s pain more effectively using ACT techniques

SUMMARY:
Background:

* Neurofibromatosis type 1 (NF1) is a genetic disorder that can cause frequent and significant pain. This pain can have a severe impact on a person s quality of life.
* Acceptance and Commitment Therapy (ACT) is a new type of therapy that may help people manage pain. It teaches behavioral techniques that can be used to change how people react to pain. ACT may help people with NF1 cope better with the pain associated with the disorder. Researchers want to test ACT techniques to see if they can improve coping in people with NF1 pain.

Objectives:

- To see if ACT can help treat chronic pain in adolescents and young adults who have NF1.

Eligibility:

- Adolescents and young adults between 12 and 21 years of age who have chronic pain associated with NF1.

Design:

* Participants will be screened with a physical exam and medical history. They will also complete a set of questionnaires about their pain levels, quality of life, and medications that they are taking.
* Participants will take part in a training workshop for ACT. It will consist of three 2-hour sessions over 2 consecutive days. The workshop will teach techniques for setting goals that reflect personal values, and changing the focus from pain avoidance to pain management. There will be practice exercises between each session.
* At the end of the workshop, participants will receive a workbook with the exercises to continue to practice at home. Participants will be encouraged to spend at least 20 minutes, three times per week, on these practice exercises.
* There will be a followup phone call to check on pain management after the workshop.
* Three months after the first study visit, participants will complete the study questionnaires again from home. They will provide more information about how they are managing their pain. The questionnaires will be returned by mail in an envelope provided by the study team.

DETAILED DESCRIPTION:
Background:

* Neurofibromatosis type 1 (NF1) is a genetic disorder that affects approximately 1 in 3,500 individuals.
* A number of common clinical manifestations, including plexiform neurofibromas, scoliosis, and chronic headaches, can cause frequent and significant pain and impact quality of life.
* Often, NF1-related pain is not well-controlled with medication and many of the medications cause significant side effects.
* To our knowledge, no studies have examined the effectiveness of behavioral interventions for chronic pain in individuals with NF1.
* Acceptance and Commitment Therapy (ACT), a newer generation of cognitive-behavioral therapy, focuses on encouraging individuals to engage in more adaptive ways of coping with pain or distress.

  * In helping individuals with pain, the goal of ACT is not to eliminate the person s pain, but to optimize the person s quality of life despite their pain.

Objectives:

* To evaluate whether the Acceptance and Commitment Therapy (ACT) group demonstrates improvement on the Modified Brief Pain Inventory scale from baseline to 3 months in adolescents and young adults with NF1 and chronic pain.
* To examine changes in patient s functional ability, quality of life, pain-related coping, pain-related anxiety, pain severity, and depression from baseline to 3 months
* To examine the effects of ACT on parents psychological well-being, overall stress, and ability to cope with their child s pain
* To explore the relationship between changes in patients pain interference, functional ability, pain-related coping, pain-related anxiety, pain severity, depression and treatment adherence with demographic variables, parent stress, and parent coping
* To collect preliminary data on the value of ACT to guide the potential development of a future phase II trial

Eligibility:

Patients ages 12 to 21 with a confirmed diagnosis of NF1.-Parents of participating patients.-The patient must indicate a score of 3 or higher on a pain item (1 5 scale) from a quality of life measure assessing the extent to which pain has interfered with the patient s daily functioning over the past month.

Design:

* This is a behavioral study to determine the feasibility and potential benefit of an ACT intervention on pain interference from baseline to 3 months post-intervention.
* A sample size of 12 patients is needed to provide 90% power for detecting a change of .77 standard deviations on the total pain interference score of the M-BPI using a 1-sided .1 level test.
* ACT workshops will be scheduled multiple times over approximately five months and will be comprised of three 2-hour sessions held over two consecutive days
* Measures assessing pain interference, pain coping, pain-related anxiety, quality of life, functional disability, depression, and pain severity will be administered to patients prior to the ACT intervention and 3 months later.
* At the same time points, a parent or legal guardian of each patient will complete measures assessing their child s quality of life, functional disability, depression, and pain severity, as well as the parent s own psychological functioning and ability to cope with their child s pain

ELIGIBILITY:
* INCLUSION CRITERIA FOR PARTICIPANT:

Subjects must be between 12 and 21 years of age at the time of the intervention. Because the research on the effectiveness of ACT with children younger than 12 is still emerging, children 11 and younger will be excluded from the present study.

For the clinical diagnosis of NF1 all study subjects must have two or more diagnostic criteria for NF1 listed below (NIH Consensus Conference):

1. Six or more cafe-au-lait spots (greater than or equal to 0.5 cm in prepubertal subjects or greater than or equal to 1.5 cm in postpuberta subjects)
2. Greater than or equal to 2 neurofibromas or 1 plexiform neurofibroma
3. Freckling in the axilla or groin
4. Optic glioma
5. Two or more Lisch nodules
6. A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
7. A first-degree relative with NF1

   Response of 3 or higher on a pain item (1 5 scale) from a self-report quality of life measure (Impact of Pediatric Illness Scale) assessing the extent to which pain has interfered with the patient s daily functioning over the past month.

   Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

   Subjects may be participating in other medical interventions for the treatment of their disease, or standard care techniques for pain management.

   No anticipated major changes in their pain regimen or enrollment on a new treatment study in the near future.

   Subjects must be able to read and comprehend the English language.

   EXCLUSION CRITERIA FOR PARTICIPANT:

   In the opinion of the PI or an AI, the subject has significant cognitive or emotional difficulties that would prevent them from being able to understand and/or participate fully in the intervention or the measures.

   Subjects who are participating in any other treatment studies, either medical or behavioral, for pain management.

   Subjects who are scheduled to begin a new drug protocol for the treatment of their NF1 during the time of their enrollment on the current study.

   Inability to travel to the NIH, for example, due to physical limitations, for the scheduled workshop and evaluations.

   No groups in regards to gender, race, or ethnicity are being excluded from participation in the trial.

   INCLUSION CRITERIA FOR PARENTS:

   Parents must have a child with NF1 who is participating in this protocol as a patient.

   Ability to read and comprehend the English language.

   Ability to understand and the willingness to sign a written informed consent document.

   If a minor patient meets all eligibility criteria but his or her parent does not (i.e., in the case where a parent does not speak English), the patient will not be allowed to participate.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-06-15; Primary Completion 2014-05-01 (Actual); Study Completion 2017-01-10 (Actual)

PRIMARY OUTCOMES:
Pain improvement | 3 months

SECONDARY OUTCOMES:
Value of the ACT for future Ph2 trial. | 6 months
Psychological well-being & stress changes in parents | 3 months
Explore improvements of pain interference, abilities, coping, anxiety,depression, etc | 3 months
Relationship between pain and treatment adherence | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Staci M Peron, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Babovic-Vuksanovic D, Widemann BC, Dombi E, Gillespie A, Wolters PL, Toledo-Tamula MA, O'Neill BP, Fox E, MacDonald T, Beck H, Packer RJ. Phase I trial of pirfenidone in children with neurofibromatosis 1 and plexiform neurofibromas. Pediatr Neurol. 2007 May;36(5):293-300. doi: 10.1016/j.pediatrneurol.2007.01.009. PMID 17509460
- [Background] Bach P, Hayes SC. The use of acceptance and commitment therapy to prevent the rehospitalization of psychotic patients: a randomized controlled trial. J Consult Clin Psychol. 2002 Oct;70(5):1129-39. doi: 10.1037//0022-006x.70.5.1129. PMID 12362963
- [Background] Blount RL, Cohen LL, Frank NC, Bachanas PJ, Smith AJ, Manimala MR, Pate JT. The Child-Adult Medical Procedure Interaction Scale-Revised: an assessment of validity. J Pediatr Psychol. 1997 Feb;22(1):73-88. doi: 10.1093/jpepsy/22.1.73. PMID 9019049